CLINICAL TRIAL: NCT02515916
Title: Fertility Preservation- Oncology Treatment Effects and Psychological Impact
Status: Terminated | Type: Observational
Why Stopped: Not enough subjects
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1301013407
Record Dates: First submitted 2015-07-09; First posted 2015-08-05 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not Interventional — This will be a prospective, non-randomized, uncontrolled study examining the effects of oncology treatments in women at risk for treatment induced ovarian failure.

SUMMARY:
The purpose of this study is assess the effects of oncology treatment on ovarian reserve and also to better understand the experiences, thoughts and feelings of women scheduled to undergo chemotherapy/radiotherapy and seeking fertility preservation at Weill Cornell Medical College (WCMC).

DETAILED DESCRIPTION:
This will be a prospective, non-randomized, uncontrolled study examining the effects of oncology treatments in women at risk for treatment induced ovarian failure. The investigators will also assess and describe the emotional, reproductive and quality of life concerns of newly diagnosed cancer patients referred for fertility preservation and determine the physical, psychosocial and quality of life differences of cancer survivors who undergo fertility preservation in comparison to those who choose not to or are unsuccessful in their attempts to cryopreserve.

Protocol Methodology:

Women who are scheduled to undergo chemotherapy and/or radiation and present for fertility preservation consultation at The Ronald O. Perelman and Claudia Cohen Center for Reproductive Medicine will be recruited for this study. All recruited patients (including those who undergo cryopreservation of embryos, eggs or ovarian tissue, those who do not undergo cryopreservation of embryos, eggs or ovarian tissue, and those who are unable to undergo cryopreservation) will be evaluated at the following time points: T1: Before starting chemotherapy initial consultation for fertility preservation; T2: Pre oncology treatment (eg chemotherapy and/or radiation; T3: At six months to 1 year post chemotherapy; Patients will subsequently have annual follow up visit for 3 years. The study involves two components: 1) Assessment of biochemical and biophysical parameters of ovarian reserve. 2) Assessment of psychosocial, reproductive and quality of life concerns of these patients

The investigators will evaluate biochemical and biophysical parameters of ovarian reserve in these patients. Anti-Müllerian hormone (AMH), follicle-stimulating hormone (FSH), estradiol (E2) levels will be drawn. In addition, the ovaries will be examined and antral follicle counts and ovarian volume will be measured on the same days that the hormone levels are drawn (if appropriate). Subjects will be asked to keep a menstrual calendar diary from baseline (pre-chemotherapy) and for 1 year post chemotherapy.

In order to assess and describe the psychosocial, reproductive and quality of life concerns of these patients, a Quality of Life (QOL) survey will be completed pre and post chemotherapy at time points:

T1: At the time of pre-chemotherapy (initial consultation for fertility preservation).

T2: Pre chemotherapy/radiation treatment. Patients who have successful cryopreservation of embryos or eggs will be asked to complete the survey on the day of embryo or egg cryopreservation or before the start date of their initial chemotherapy treatment. Patients who do not have successful cryopreservation of embryos or eggs will be asked to complete the survey after receiving notification that the fertility preservation treatment is cancelled. Patients who do not choose to cryopreserve embryos or eggs will be asked to fill out the survey before the start date of their initial chemotherapy treatment. Participants will be mailed or given a survey instrument and the data collected either in person, by mail, or by telephone.

T3: At six months to 1 year post chemotherapy, patients will be asked to complete the final survey by phone or by mail. Systematic reminders (mail and phone) will be used to ensure return of the surveys. Each study survey should take approximately 40-55 minutes to complete. The domains assessed will include psychological functioning, reproductive and fertility preservation concerns, relationship satisfaction, and quality of life prior to and following potential fertility preservation and initial chemotherapy treatment for breast cancer. Participants do not have to respond to any question that they choose not to answer.

Study Instruments: Quality of Life (QOL) survey-

1. Psychosocial History and Background Information Form
2. Symptom Checklist (SCL)
3. Center for Epidemiologic Studies-Depression (CES-D)
4. Dyadic Adjustment Scale (DAS)
5. The Reproductive Concerns Scale (RCS)
6. Impact of Events Scale (IES)
7. The Life Orientation Test (LOT-R)
8. The Functional Assessment of Cancer Therapy-General

Data will be collected and analyzed. This new data will help us establish a better understanding of the effects of chemotherapy on total ovarian reserve and assist clinicians caring for patients of reproductive age in counseling these patients. The findings of study will also bring attention to the understudied area of fertility preservation and cancer survivorship. The investigators propose that by studying the short and long-term psychosocial impact of fertility preservation with comparison between those who undergo cryopreservation with those who do not, the investigators will be able to assess if psychosocial changes occur over time and identify points for future intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-45
* Women seeking fertility preservation at WCMC
* Women who will undergo oncology treatments that will likely cause reduced fertility potential.

Exclusion Criteria:

* Women who do not meet the inclusion criteria

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women scheduled to undergo chemotherpay/radiotherapy and are seeking fertility preservation at WCMC
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
AMH (anti-mullerian hormone) blood levels | Up to 3 years
  To determine if fertility reserve is affected by oncology treatment.
Quality of life on the Dyadic Adjustment Scale | 3 years
  To determine if there is any psychological impact of oncology treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Schattman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Ronald O. Perelmand and Claudia Cohen Center for Reproductive Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No